CLINICAL TRIAL: NCT04900467
Title: Multicenter, Randomized, Open-label Trial Comparing the Immunological Efficacy of a Vaccine Regimen Combining Two Covid19 mRNA Vaccines (Pfizer-BioNTech and Moderna) With That of a Homologous Vaccination of Each Covid19 mRNA Vaccine: Non-inferiority Trial
Brief Title: Compare Immunological Efficacy of a Vaccine Regimen Combining Two Covid19 mRNA Vaccines (Pfizer-BioNTech and Moderna) With That of a Homologous Vaccination of Each Covid19 mRNA Vaccine
Acronym: ARNCOMBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: COVIREIVAC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP210605; 2021-002174-52 (EudraCT Number)
Record Dates: First submitted 2021-05-21; First posted 2021-05-25 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Adult Who Received a First Dose of an mRNA Vaccine (Pfizer-BioNTech or Moderna) and Need to Receive a Second Dose
Keywords: COVID 19; mRNA vaccines; Immunology; mRNA-1273; BNT162b2
MeSH Terms: conditions — COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pfizer-Pfizer (Active Comparator): Pfizer-Pfizer Length of use : 1 day
  Interventions: Biological: Pfizer
- Pfizer-Moderna (Experimental): Pfizer-Moderna Length of use : 1 day
  Interventions: Biological: Pfizer; Biological: Moderna
- Moderna- Moderna (Active Comparator): Moderna- Moderna Length of use : 1 day
  Interventions: Biological: Moderna
- Moderna - Pfizer (Experimental): Moderna - Pfizer Length of use : 1 day
  Interventions: Biological: Pfizer; Biological: Moderna

INTERVENTIONS:
Biological: Pfizer — BNT162b2 (Comirnaty®), Pfizer/BioNTech, mARN vaccine,
  Arms: Moderna - Pfizer; Pfizer-Moderna; Pfizer-Pfizer
Biological: Moderna — mRNA-1273, COVID-19 Vaccine Moderna, mARN vaccine, administrated by intramuscular
  Arms: Moderna - Pfizer; Moderna- Moderna; Pfizer-Moderna

SUMMARY:
As part of the COVID 19 vaccine campaign, the two mRNA vaccines, BNT162b2 (COMIRNATY®) and mRNA-1273 COVID-19 vaccine Moderna, are administered in two doses in subjects without a history of SARS-CoV-2 infection . In accordance with the marketing authorization for vaccines, HAS recommends that subjects who have received one dose of an mRNA vaccine receive a second dose of the same vaccine with an interval between the 2 doses of 4 to 6 weeks. These two vaccines are based on very similar technologies but were developed independently. Given the similarities between these two vaccines, the choice between the two, for the moment, is based solely on the availability of doses and on logistical constraints. Since April 14, the interval between the two doses of the mRNA vaccines is 42 days.

WHO has announced that in the absence of available data, vaccine interchangeability cannot be recommended. However, to facilitate the organization of the vaccination campaign and allow faster vaccination of the population, it would be desirable to be able to use either one or the other mRNA vaccine for the 2nd dose.

In order to be able to recommend the interchangeability of the 2 mRNA vaccines, it is proposed to evaluate the immunogenicity of a scheme combining the two Covid 19 mRNA vaccines (i.e. a 2nd dose of vaccine with the Moderna vaccine after a first dose of the Pfizer vaccine or 2nd dose of Pfizer vaccine after a first dose of Moderna vaccine) compared to that of a standard vaccination schedule with two doses of the same Covid 19 mRNA vaccine.

DETAILED DESCRIPTION:
Covid 19 has infected more than 132 million people around the world (https://covid19.who.int/, data from 04/07/21). In record time, effective vaccines were developed allowing the start of the vaccination campaign less than a year after the outbreak was declared by WHO.

To date, more than 604 million vaccine doses have been administered worldwide (https://covid19.who.int/, data from 04/07/21).

On December 21, 2020, the first mRNA vaccine developed by Pfizer and BioNTech obtained a marketing authorization (conditional AMM) in Europe for the active immunization of people 16 years of age and over to prevent Covid-19 due to SARS -CoV-2. Then, on January 6, 2021 Moderna in turn obtained a conditional Marketing Authorization for the indication of active immunization to prevent Covid-19 due to SARS-CoV-2 in subjects 18 years of age and over.

In France, more than 7 million injections have been performed with the Pfizer / BioNTech vaccine and more than 617,000 doses of the Moderna vaccine.

The two mRNA vaccines, BNT162b2 (COMIRNATY®) from Pfizer / BioNTech and mRNA-1273 COVID-19 vaccine Moderna, are given on a two-dose schedule in subjects without a history of SARS-CoV-2 infection. In accordance with the AMM for vaccines, HAS recommends that subjects who have received one dose of an mRNA vaccine receive a second dose of the same vaccine. The recommended interval between the 2 doses is 4 to 6 weeks. These two vaccines are based on very similar technologies but were developed independently. Given the similarities between these two vaccines, the choice between the two, for the moment, is based solely on the availability of doses and on logistical constraints.

Since 14 April, the interval between the two doses of mRNA vaccines is 42 days. In order to facilitate the organisation of the vaccination campaign and to enable the population to be vaccinated more quickly, it would seem desirable to be able to use either COVID 19 RNA vaccine for the 2nd vaccine dose. However, the WHO has announced that, in the absence of available data, the interchangeability of vaccines cannot be recommended.

In order to be able to recommend the interchangeability of the 2 mRNA vaccines, the ARN Combi trial aims to compare the immunogenicity of a standard vaccine regimen (second dose of the same Covid 19 mRNA vaccine) to that of a regimen combining the two Covid 19 mRNA vaccines (i.e. either a 2nd dose of vaccine with Moderna vaccine after a first dose of Pfizer vaccine or a 2nd dose of Pfizer vaccine after a first dose of Moderna vaccine)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Having received a first dose of one of the two mRNA vaccines (Pfizer-BioNTech or Moderna) as recommended.
3. For whom a 2nd dose of mRNA vaccine is planned within 4 to 6 weeks (according to the recommendations of the HAS and the ANSM).
4. Without a history of SARS-CoV-2 infection (negative PCR, negative antigen test or negative chest CT or SARS-CoV-2 serology)
5. Healthy or in stable health if pre-existing medical history. Stable health is defined as an existing disease that has not required a significant change in treatment or hospitalisation for worsening in the 3 months prior to inclusion, and for which neither a significant change in treatment or hospitalisation for worsening of the disease is envisaged in the near future
6. Able to understand and comply with the research procedures as judged by the investigator
7. Informed consent signed by the participant and the investigator.
8. Person affiliated to a social security scheme.

Exclusion Criteria:

1. History of SARS-CoV-2 infection at the inclusion visit or between the 2 vaccine doses (documented by positive PCR, positive antigen test or positive chest CT or positive SARS-CoV-2 serology.
2. Acute febrile infection (body temperature ≥ 38.0°C) within the previous 72 hours and/or with symptoms suggestive of COVID-19 or case contact within the last 14 days prior to the inclusion visit. Sick or febrile subjects may be re-invited for a new inclusion visit during the inclusion period when they no longer have these symptoms)
3. Immunosuppressive medications such as corticosteroids at a dosage > 10 mg prednisone equivalent/day (excluding topical preparations and inhalers) within 3 months prior to inclusion or within 6 months for chemotherapy.
4. Treatment with immunoglobulin or other blood product within 3 months prior to inclusion or with planned administration of immunoglobulin or blood product before the end of the study.
5. Known HIV, HCV or HBV infection.
6. Any immunosuppressive condition, such as cancer, that may reduce the immune response.
7. The use of experimental Ig, experimental monoclonal antibodies or convalescent serum is not permitted during the study.
8. Pregnant or breastfeeding.
9. Participation in any other research involving humans (Jardé 1 or Jardé 2) within 4 weeks prior to the inclusion visit
10. Person subject to a legal protection measure (guardianship, curatorship or safeguard measure).
11. History of severe adverse reactions after vaccine administration including anaphylactic reaction and associated symptoms such as rash, difficulty breathing, angiodema and abdominal pain, or a history of allergic reaction that may be exacerbated by a component of the SARS-COV-2 vaccine at the time of the first vaccine injection
12. Participant who has been vaccinated against BCG in the previous year.
13. Having received a vaccination within 4 weeks prior to the first injection or scheduled to receive a licensed vaccine 4 weeks after the last injection.
14. History of severe allergic manifestations
15. Any bleeding disorder considered to be a contraindication to intramuscular injection or having had a phlebotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Anti-Spike IgG titer | 28 days
  Anti-Spike IgG titer measured by ELISA and neutralising antibodies to European SARS-CoV-2 and SARS-CoV-2 variants 28 days after the second injection.

SECONDARY OUTCOMES:
Adverse events | 6 months
  Any adverse events, local and systemic reactions occurring up to 180 days (6 months) after the second injection.

CONTACTS AND LOCATIONS:
Overall Officials: Odile LAUNAY, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Cécile JANSSEN, Principal Investigator — Centre Hospitalier Annecy Genevois
Locations (1):
- CIC 1417 Cochin-Pasteur, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Janssen C, Cachanado M, Ninove L, Lachatre M, Michon J, Epaulard O, Maakaroun-Vermesse Z, Chidiac C, Laviolle B, Aumaitre H, Assaf A, Lacombe K, Schmidt-Mutter C, Botelho-Nevers E, Briere M, Boisson T, Loubet P, Bienvenu B, Bouchaud O, Touati A, Pereira C, Rousseau A, Berard L, Montil M, de Lamballerie X, Simon T, Launay O; ARNCOMBI Study Group. Immunogenicity and reactogenicity of heterologous and homologous mRNA-1273 and BNT162b2 vaccination: A multicenter non-inferiority randomized trial. EClinicalMedicine. 2022 Jun;48:101444. doi: 10.1016/j.eclinm.2022.101444. Epub 2022 May 12. PMID 35582124